CLINICAL TRIAL: NCT05323006
Title: The Effect of the Scapular Stabilization Exercises on the Clavicular Movement on the Girl Adolescents,
Brief Title: Scapular Stabilization Exercises on the Clavicular Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaziantep Islam Science and Technology University (Other)
Responsible Party: Principal Investigator, Gönül Elpeze, Physiotherapist, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: HKU-GE-Clavicular movement
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Clavicle
Keywords: adolescent,; clavicula,; scapula,; exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scapular stabilization exercises (Active Comparator): the effect of the scapular stabilization exercises on clavicular movement
  Interventions: Other: scapular stabilization exercises
- no intervention (No Intervention): no intervention

INTERVENTIONS:
Other: scapular stabilization exercises — the effect of the scapular stabilization exercise on the clavicular motion on the adolescent girls
  Arms: scapular stabilization exercises

SUMMARY:
This study was planned to indicate efficiacy of the scapular stabilization exercises on the clavicula movements.

DETAILED DESCRIPTION:
All subjects in the study were evaluated for range of motion (Goniometer), muscle strength (Manuel Muscle Strength Test), angular displacements of clavicula during abduction and skapular plan elevation of arm (Video Analysis Method), disability of the arm (Quıck Dash Turkish). The study was applied in two groups for three times per week during 8 weeeks.

ELIGIBILITY:
Inclusion Criteria:

* Having no ınjury for lower anda upper extremites

Exclusion Criteria:

* Having ınjury for lower anda upper extremites

Ages: 10 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2017-07-11 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
the effect of the scapular stabilization exercises | 1 Year
  clavicular elevation and depression

CONTACTS AND LOCATIONS:
Overall Officials: GÖNÜL ELPEZE, Principal Investigator — HKU
Locations (1):
- Hasan Kalyoncu Üniversitesi, Şehitkamil, Gazi̇antep, Turkey (Türkiye)